CLINICAL TRIAL: NCT06269536
Title: A Study on Therapeutic Potential of Stress-reducing Intervention in Patients With Urothelial Carcinoma
Brief Title: Stress-reducing Intervention in Urothelial Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UC-SK004
Record Dates: First submitted 2024-01-17; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Bladder Cancer
Keywords: Muscle-Infiltrating Urothelial Carcinoma; Neoadjuvant Chemotherapy; Standard of Care; Heart-Rate Variability; Biofeedback Intervention; Inflammation; Quality of Life; Cognitive Functions; Salivary Cortisol Slopes; Circadian Rhythms; Sleep Quality
MeSH Terms: conditions — Urinary Bladder Neoplasms; Inflammation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart-rate variability (HRV) biofeedback intervention + standard of care (Experimental): Deep paced breathing with the HRV monitoring performed three times a day for seven minutes during three months with standard of care.
  Interventions: Other: HRV biofeedback
- Standard of care (No Intervention): Gemcitabine 1000 mg/m2 + Cisplatin 70 mg/m2 day 1 (new course day 22) or Methotrexate 30 mg/m2 day 1, Doxorubicin 30 mg/m2 day 2, Vinblastine 3 mg/m2 day 2, Cisplatin 70 mg/m2 day 2 with Pegfilgrastim 6 mg s.c. day 4 (new course day 15) up to 4 courses followed by radical cystectomy or irradiation with cisplatin 70 mg/m2 weekly.

INTERVENTIONS:
Other: HRV biofeedback — Daily deep paced breathing 3-times (minimum 7 minutes each) for 3 months
  Other Names: physiologic
  Arms: Heart-rate variability (HRV) biofeedback intervention + standard of care

SUMMARY:
The aim of this interventional study is to test the heart-rate variability biofeedback intervention (HRV BI) in patients with muscle-infiltrating bladder carcinoma (MIBC) treated with chemotherapy based on cisplatin in neoadjuvant setting followed by local therapy (standard of care, SOC) compared to SOC alone.

DETAILED DESCRIPTION:
This is a prospective, interventional, clinical study with a target of 50 subjects and an anticipated total duration of 36 months.

The goal of this study is to test the HRV BI in patients with MIBC treated with total of 3 to 4 courses of chemotherapy Gemcitabine 1000 mg/m2 + Cisplatin 70 mg/m2 day 1 (GC, new course day 22) or Methotrexate 30 mg/m2 day 1, Doxorubicin 30 mg/m2 day 2, Vinblastine 3 mg/m2 day 2, Cisplatin 70 mg/m2 day 2 with Pegfilgrastim 6 mg s.c. day 4 (ddMVAC, new course day 15) in neoadjuvant setting followed by radical cystectomy or irradiation concomitantly with cisplatin 70 mg/m2 weekly (SOC) and compare to SOC.

Participants will undergo 4 sessions of HRV BI with the trainer where they will learn about the prognostic role of the vagal nerve in cancer and in reducing distress and pain, and how to perform deep paced breathing with the HRV monitoring. They will perform the training daily (3-times, minimum 7 minutes each) at home with the online control for 3 months.

Researchers will compare the effect of addition of 3-months training of HRV BI to SOC on inflammation, HRV, quality of life (QoL), cognitive functions, salivary cortisol slopes, sleep quality and treatment outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Patients older than 18 years.
2. Evidence of muscle-infiltrating urothelial bladder carcinoma (including variants) by biopsy.
3. No prior chemotherapy.
4. No previous malignancy, except for basal-cell carcinoma of the skin within last 5 years.
5. Adequate renal functions: measured or calculated (by Cockcroft formula) creatinine clearance > 60 ml/min.
6. Absolute granulocytes count 1,500/mm3 or higher, platelets 100,000/mm3 or higher, bilirubin 1.5x the upper limit of normal value and lower.
7. Adequate liver functions.
8. Basic computer skills.
9. Signed informed consent.

Exclusion criteria:

1. Diabetes mellitus with symptomatic neuropathy.
2. Using antiarrhythmic drugs, opiates and/or antidepressants.
3. Implanted permanent pacemaker (PPM).
4. Human Immunodeficiency Virus (HIV) infection.
5. Not fitting inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Primary Objective: Inflammation | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on inflammation (IL-6, Tumor necrosis factor α, IL-10 in pg/ml).
Primary Objective: Heart Rate Variability (HRV) | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on HRV indexed by the root mean square of successive differences between heartbeats (RMSSD) in ms.
Primary Objective: Quality of Life (QoL) | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on EORTC-QLQ-C30 (version 3) score. The EORTC-QLQ-C30 has 30 items divided into five functional scales (physical, role, cognitive, emotional, and social), and three symptom scales (fatigue, pain, and nausea and vomiting). The score for each scale as well as the sum score for the whole instrument is standardized to values 0 to 100, with a higher score meaning a worse outcome.
Primary Objective: Working memory | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on working memory measured by digit span test score (the number of remembered digits in the longest passed sequence), for both forward and backward condition.
Primary objective: Executive function | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on executive function measured by Stroop task mean response time for color-word condition.
Primary objective: Salivary Cortisol Slopes | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on salivary cortisol slopes (difference between bedtime and awakening saliva cortisol concentration in ng/ml).
Primary objective: Sleep Quality | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on sleep quality measured by both actigraphy and self-report data. The main variables are total time spent sleeping (in hours and minutes), and sleep efficiency (proportion of time spent sleeping vs. time spent in bed trying to sleep).

SECONDARY OUTCOMES:
Secondary objective: Serious Adverse Events | 36 months
  The effect of 3-months heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on serious adverse events (SAEs) of chemotherapy.
Secondary objective: Disease-Free Survival (DFS) | 60 months
  The effect of 3-months heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on disease-free survival (DFS).
Secondary objective: Overall Survival (OS) | 60 months
  The effect of 3-months heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Palacka, Principal Investigator — Faculty of Medicine, Comenius University in Bratislava
Locations (1):
- National Cancer Institute, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data of HRV, cognitive functions, quality of life, inflammatory markers, salivary cortisol, sleep quality, physical activity and psychological questionnaires.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will became available together with the publication and will be available for 5 years.
Access Criteria: Open.